CLINICAL TRIAL: NCT04727983
Title: Effects of External Neuromuscular Electrical Stimulation in Women With Urgency Urinary Incontinence: A Randomized Sham-Controlled Study
Brief Title: Effects of External Neuromuscular Electrical Stimulation in Women With Urgency Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, TUĞBA BİRBEN, Tugba Birben, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/07 decision, 21 protocol
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Physiotherapy; Women's Health; Urge Incontinence; Electrical Stimulation
Keywords: Urge urinary incontinence; Electrical stimulation; Neuromuscular electrical stimulation (NMES); Physiotherapy
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 2 groups randomly.
Who Masked: Participant
Masking Description: This study was planned single blinded randomized control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Pelvic Floor Muscle Function (No Intervention): Pelvic floor muscle function will be evulated with the Modified Oxford Scale
- Bladder function (No Intervention): Bladder function will be evulated with the urinary diary for 3 days
- Incontinence Symptoms (No Intervention): Incontinence Symptoms will be evulated with The International Incontinence Consultation Questionnaire-Short Form (ICIQ-SF) and the Coital Incontinence Score (CIS)
- Quality of Life (No Intervention): Quality of life will be evulated with the King Health Questionnaire (KHQ)
- Sexual Function (No Intervention): Sexual Function will be evaluated with Pelvic Organ Prolapse / Urinary Incontinence Sexual Questionnaire (PISQ-12).
- NMES group (Experimental): The first group will be given Neuromuscular Electrical Stimulation (NMES) and lifestyle suggestions (LSS)
  Interventions: Device: Electrotherapy
- SHAM ES group (Sham Comparator): The second group will be given sham NMES in addition to LSS
  Interventions: Device: Sham Electrotherapy
- End of Treatment Special Evaluations (No Intervention): Subjective perception of improvement and treatment satisfaction of the patients will be questioned

INTERVENTIONS:
Device: Electrotherapy — The first group will be given Neuromuscular Electrical Stimulation (NMES) and lifestyle suggestions (LSS) (NMES group)
  Arms: NMES group
Device: Sham Electrotherapy — The second group will be given sham NMES in addition to LSS (SHAM ES group)
  Arms: SHAM ES group

SUMMARY:
To reveal the effects of Neuromuscular Electrical Stimulation (NMES) applied over the thigh on incontinence symptoms, pelvic floor muscle function, bladder function, quality of life and sexual function in women with urge urinary incontinence (UUI) symptoms. Our goal is to contribute to the literature on electrical stimulation (ES) applications used in UUI treatment.

Female patients aged 18-65 years with UUI symptoms will be included in the study. Patients will be divided into 2 groups randomly. The first group will be given Neuromuscular Electrical Stimulation (NMES) and lifestyle suggestions (LSS) (NMES group). The second group will be given sham NMES in addition to LSS (SHAM ES group). Information about bladder irritants, voiding posture and behavior, weight control and pelvic floor muscle training will be provided in the LSS. ES applications will be performed 3 days a week for 30 minutes per session for 8 weeks. All participants will be evaluated pretreatment, after the 4th week and posttreatment. Pelvic floor muscle function will evulate with the Modified Oxford Scale. In addition, women's bladder function with the urinary diary for 3 days, incontinence symptoms with the International Incontinence Consultation Questionnaire-Short Form (ICIQ-SF) and the Coital Incontinence Score (CIS), quality of life with the King Health Questionnaire (KHQ) and Sexual Function will be evaluated with Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). At the end of the 8th week, both the Subjective perception of improvement and treatment satisfaction of the patients will be questioned

DETAILED DESCRIPTION:
Our study will be carried out with female patients between the ages of 18-65 who have Urge urinary Incontinence (UUI) symptoms and applied to the Recep Tayyip Erdogan University Training and Research Hospital, Gynecology and Obstetrics Policlinic. Inclusion criterias are; who do not want to use medication, who do not benefit from medication for a long time or who do not use any medication. Exclusion criterias are; Those with any malignant conditions, those with neurological disease, those with infection, pregnant women, those with pelvic organ prolapse above stage 2 according to the POP-Q staging, those with cardiac implants and pacemakers, those with cardiac arrhythmia, those with urinary retention, those with sensory loss, copper coil intrauterine those who wear a vehicle, patients with metal implants and patients with communication and cooperation problems.

Before starting the study, all participants will be questioned about demographic and physical characteristics, medical, obstetric, gynecological and urological history and drug use. After these evaluations, sensory and reflex evaluations will be made. Sensory assessment will be performed with a light touch test to the hip circumference and pelvic floor muscles. In reflex evaluation, anal and bulbocavernous reflexes will be checked. All of the applications will be carried out by Specialist Physiotherapist Tuğba Birben under the supervision of Specialist Gynecologist Physician Beril Gürlek.

Our study will be in 2 groups. It is estimated that the number of people will consist of 40 volunteers, with 20 patients for each group. The sample size will be determined after the pilot study. Patients who were diagnosed with UUI, met the study criteria and accepted to be included in the study, within a period of 9 months after the approval of the ethics committee, with the four-block randomization method, via the website https://www.sealedenvelope.com/simple-randomiser/v1/lists will be included in groups according to randomization. lifestyle suggestions (LSS)+ NMES (NMES group) will be applied to the first group and LSS + SHAM Electrical Stimulation (SHAM ES group) will be applied to the second group. Each group will be included in the 8-week treatment program for 30 minutes, 3 days a week.

Pelvic floor muscle function of all participants will be evaluated with the Modified Oxford Scale before treatment, at the end of the 4th week and after treatment. In addition, women's bladder function with the urinary diary, incontinence symptoms with the International Incontinence Consultation Questionnaire-Short Form (ICIQ-SF) and the Coital Incontinence Score (CIS), quality of life with the King Health Questionnaire (KHQ) and Sexual Function will be evaluated with Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). At the end of the 8th week, both the Subjective perception of improvement and treatment satisfaction of the patients will be questioned.

ELIGIBILITY:
Inclusion Criteria:

* who do not want to use medication,
* who do not benefit from medication for a long time
* who do not use any medication

Exclusion Criteria:

* Those with any malignant conditions,
* those with neurological disease,
* those with infection,
* pregnancy,
* those with pelvic organ prolapse above stage 2 according to the POP-Q staging,
* those with cardiac implants and pacemakers,
* those with cardiac arrhythmia,
* those with urinary retention,
* those with sensory loss,
* copper coil intrauterine those who wear a vehicle,
* patients with metal implants
* patients with communication and cooperation problems

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients aged 18-65 years with UUI symptoms will be included in the study.
Enrollment: 34 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Function | 8 weeks
  Pelvic Floor Muscle Function will be evulated with The Modified Oxford Scale (MOS).
  It rates the Pelvic floor muscle contraction on a scale of 0-5; 0 = no contraction; 1 = minor muscle 'flicker'; 2 = weak muscle contraction; 3 = moderate muscle contraction; 4 = good muscle contraction and 5 = strong muscle contraction.
Bladder Function | 8 weeks
  Bladder Function will be evulated with the bladder diary for 3 days
Incontinence Symptoms | 8 weeks
  Incontinence symptoms will be evulated with The International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF) it has 5 questions and total score ranges is 1 - 5 (slight), 6 - 12 (moderate), 13 - 18 (severe) and 19 - 21 (very severe).
Quality of Life Questionnaire | 8 weeks
  quality of life will be evulated with the King's Health Questionnaire (KHQ) It consists of 3 parts. In the first part; 2 questions evaluating General health perception, in the second part; 19 questions that divide the quality of life into different areas (Incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/ energy, general health status, symptom severity) and in the third part; It consists of 11 questions evaluating the severity of urinary symptoms.
  The individual items in the domains are scaled from 0 (best) to 100 worst. Another dimension is added which is called as Symptom severity scale; where in there are 10 different bladder symptoms, the score ranges from 0 to 30 and the values are not converted to percentages.
Sexual Function | 8 weeks
  Sexual Function will be evulated with the Pelvic Organ Prolapse Urinary Incontinence Sexual Questionnaire - 12 (Short Form) (PISQ-12-SF) The questionnaire is based on 12 items that allow investigation of three different domains of sexual life; behavior (items 1-4), physical (items 5-9) and partner-related (items 10-12). Scores are calculated by totaling the scores for each question with 0 = always to 4 = never. Reversed scoring is used for items 1, 2, 3 and 4. Higher PISQ-12-SF scores indicate a better sexual function. Maximum score is 48.
End of Treatment Special Evaluations | 8 weeks
  Subjective perception of improvement and treatment satisfaction of the patients will be questioned

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA BIRBEN, MSc, Study Director — Recep Tayyıp Erdogan University Guneysu Vocational School of Physical Therapy and Rehabilitation
Locations (1):
- Recep Tayyıp Erdogan University Guneysu Vocational School of Physical Therapy and Rehabilitation, Rize, Guneysu, Turkey (Türkiye)

REFERENCES:
- [Derived] Kurt TB, Yilmaz B, Celenay ST. Effects of external neuromuscular electrical stimulation in women with urgency urinary incontinence: a randomized sham-controlled study. World J Urol. 2024 Jul 21;42(1):423. doi: 10.1007/s00345-024-05126-7. PMID 39033475